CLINICAL TRIAL: NCT05662189
Title: Assessment of Pancreatic Beta Cell Mass and Function with the Aid of Positron Emission Tomography Imaging in Human Diabetes Mellitus
Brief Title: Assessment of Pancreatic Beta Cell Mass and Function by Positron Emission Tomography Imaging in Human Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: University of Parma (Other)
Responsible Party: Principal Investigator, Riccardo Bonadonna, Prof, Azienda Ospedaliero-Universitaria di Parma
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 462
Record Dates: First submitted 2022-12-01; First posted 2022-12-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Type1diabetes; Type2diabetes; Pre Diabetes; Hyperinsulinism
Keywords: diabetes; beta-cell; exendin; PET-CT
MeSH Terms: conditions — Glucose Intolerance; Hyperinsulinism; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Obese people with normal glucose regulation , patients with long standing or newly diagnosed type 1 diabetes, patients with long standing or newly diagnosed type 2 diabetes, subjects with pre-diabetes, and lean healthy age- and gender-matched controls will participate in two study sessions on two separate days:
  * Session A (Endocrinology and Metabolic Diseases Unit) - Quantitation of beta cell functional mass (BCFxM) by mixed-meal test
  * Session B (Nuclear Medicine Unit) - Quantitation of beta cell mass (BCM) by PET-CT scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- long standing type 1 diabetes (> 20 yrs) (Other): 68Ga-exendin4 PET-CT scan +mixed meal test
  Interventions: Drug: 68Ga-exendin-4; Other: mixed meal test
- newly diagnosed type 1 diabetes (< 5yrs) (Other): 68Ga-exendin4 PET-CT scan +mixed meal test
  Interventions: Drug: 68Ga-exendin-4; Other: mixed meal test
- long standing type 2 diabetes (> 20 yrs) (Other): 68Ga-exendin4 PET-CT scan +mixed meal test
  Interventions: Drug: 68Ga-exendin-4; Other: mixed meal test
- newly diagnosed type 2 diabetes (<6 months) (Other): 68Ga-exendin4 PET-CT scan +mixed meal test
  Interventions: Drug: 68Ga-exendin-4; Other: mixed meal test
- pre-diabetes (Other): 68Ga-exendin4 PET-CT scan +mixed meal test
  Interventions: Drug: 68Ga-exendin-4; Other: mixed meal test
- hyperinsulinemic (Other): 68Ga-exendin4 PET-CT scan +mixed meal test
  Interventions: Drug: 68Ga-exendin-4; Other: mixed meal test
- control (Other): 68Ga-exendin4 PET-CT scan +mixed meal test
  Interventions: Drug: 68Ga-exendin-4; Other: mixed meal test

INTERVENTIONS:
Drug: 68Ga-exendin-4 — 68Ga-exendin4 PET-CT scan
Other: mixed meal test — before and after a standardized mixed meal venous blood samples will be collected at time intervals to measure plasma glucose, C-peptide,insulin, glucagon, glucagon-like peptide 1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP) curves

SUMMARY:
The goals of this project are to build an experimental tool to dissect out in vivo pancreatic beta cell mass (BCM) and beta cell function (BCF) and to assess for the first time these two determinants of beta cell functional mass (BCFxM) in obesity and in various stages of type 1 and type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Pancreatic beta cell functional mass (BCFxM) can be loosely defined as the product of beta cell mass (BCM) multiplied by beta cell function (BCF). Current in vivo methods (e.g. hyperglycemic clamp, intravenous glucose tolerance test, oral glucose tolerance test, mixed meal tolerance test) actually assess BCFxM, not beta cell function per se. Loss of BCFxM is at the heart of the etiology and pathogenesis of both type 1 (2) and type 2 diabetes mellitus. In the former, destruction of beta cell mass by autoimmune insulitis is the the primary determinant of BCFxM loss. In the latter, beta cell mass loss is about 25-35% and keeps increasing with the duration of the disease, but an additional key role is played by the loss of beta cell function. Previous dogma held that in type 1 diabetes complete destruction of beta cells was achieved within ≈5 years from diagnosis. Recent data have challenged this concept and shown that residues of both beta cells and BCFxM (i.e. nutrient-stimulated C-peptide secretion, which is equimolar and simultaneous to insulin secretion and is a much better biomarker of BCFxM than insulin concentration) are detectable even decades after diagnosis. Exendin-4 has been already labeled with a positron emitting nuclide and made amenable to PET imaging for diagnostic purposes. Under rigorous experimental conditions, beta cell standardized uptake per volume (SUV) of the ligand could be assessed. Furthermore, current PET-CT instruments can also provide a measure of pancreatic volume BCFxM can be determined accurately by mathematical modeling of relatively simple tests, such as a mixed meal.

The investigators will assess the relative roles of beta cell mass (BCM) and beta cell function (BCF) in two polar BCFxM groups : people with long-standing type 1 diabetes (close to 0 BCFxM) and obese people with normal glucose regulation (highest expected BCFxM), i.e. the investigators will test our method in a negative control (type 1 diabetes) and in a strongly positive control (uncomplicated obesity). A group of lean controls will be studied to ascertain that their BCMs, as determined by 68GA-exendin-4 PET-CT, fall, as they should, in the intermediate range between type 1 diabetes and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years; ≤ 75 years
* Both sexes
* Good health
* Absence of exclusion criteria
* Able to understand methods, goals, and implications of the research and of delivering a free, written informed consent

Exclusion Criteria:

* Hemoglobin < 12 g/dl
* HbA1c > 10%
* Pregnancy or breast-feeding
* If not in menopause, women not using effective birth control methods or not willing to undergo a pregnancy test
* History of severe psychiatric disorder or alcohol abuse
* Recent head traumas (<6 months)
* Active neurologic diseases
* Claustrophobia
* Active malignant neoplasms
* Severe kidney and/or liver disease
* Recent (<6 months) major adverse cardiovascular events
* Heart failure (class NYHA 3-4)
* Drugs known to affect beta cell function and/or insulin sensitivity
* Current or past treatment with GLP1R-agonists
* Intolerance to exenatide
* Endocrine diseases, other than diabetes mellitus, known to affect beta cell function and/or insulin sensitivity, except well controlled hypothyroidism or adrenal insufficiency
* COPD on day time oxygen therapy
* Any current acute disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
BCF x M | through study completion, an average of 3 months after enrolment
  BCFxM=parameters derived from mixed meal test
  Beta cell function(BCF)=BCFxM/BCM
pancreatic beta cell mass (BCM) | through study completion, an average of 3 months after enrolment
  Beta cell mass index (BCM) = 68GA-exendin-4 Standard Uptake Value (SUV)*pancreatic volume
pancreatic beta cell function (BCF) | through study completion, an average of 3 months after enrolment
  BCFxM/BCM

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Bonadonna, MD, Principal Investigator — Azienda Ospedaliero Universitaria di Parma, University of Parma
Locations (1):
- Azienda Ospedaliero Universitaria di Parma, Parma, Pr, Italy